CLINICAL TRIAL: NCT03569748
Title: Randomized, Non-Inferiority Trial ComparingCigarette Consumption, Adoption Rates, Acceptability, Tolerability, and Tobacco Harm Reduction Potential in Smokers Switching to Heated Tobacco Products or Electronic Cigarettes: Study Protocol
Brief Title: Heated Tobacco Products vs Electronic Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Collaborators: Philip Morris Products S.A. (Industry)
Responsible Party: Principal Investigator, Enrico Gian Maria Mondati, Researcher of Internal Medicine, University of Catania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 215/2017/PO
Record Dates: First submitted 2018-05-14; First posted 2018-06-26 (Actual); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Smoking, Cigarette
Keywords: smoking; harm reduction; electronic cigarette; heated tobacco product
MeSH Terms: conditions — Cigarette Smoking; Smoking; Harm Reduction; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IQOS (Experimental): HEAT NOT BURN REDUCED RISK PRODUCT
  Interventions: Device: IQOS
- E-CIG (Active Comparator): ELECTRONIC CIGARETTE REDUCED RISK PRODUCT
  Interventions: Device: E-CIG

INTERVENTIONS:
Device: IQOS — IQOS USE FOR 12 WEEKS
  Arms: IQOS
Device: E-CIG — ELECTRONIC CIGARETTE FOR 12 WEEKS
  Arms: E-CIG

SUMMARY:
This is a 12-weeks, open label, non-inferiority trial comparing HTPs vs ECs in terms of efficacy, adoption rate and acceptability, tolerability, and tobacco harm reduction in 220 healthy smokers, not motivated to quit, randomized (1:1) to switch to one of these products. The duration of the study, from the enrollment to the study close out for all the patients at week 24 (follow-up), will be approximately 12 months. Enrollment period will last about 6 months with the support of a multi-channel advertising method. This will include location-based advertising on social networks, advertising in local media, information days organized within the city.

DETAILED DESCRIPTION:
Before the baseline visit, a face to face screening (V0) for pre-eligibility checks will be conducted. Subjects will be asked to practice with the step test for 10-15 minand will be instructed how to collect and store their morning urine before bringing it to the hospital on their Baseline visit (V1). This study will consist of a baseline visit (V1) and 6 follow-up study visits (V2-V7). At baseline (V1), participants will be randomized in two separate study groups. The randomization sequence will be computer generated by using blocks size of 5, with an allocation ratio of 1:1 for each of the study products (IQOS, JustFog-EC). Subjects will use and familiarize with their allocated product, as per randomization. They will be trained and counseled on the use of their allocated study product; oral explanation and practical demonstration will be followed by product trial during which participants will also have the option to try and choose their preferred flavour (either from a selection of 3 e-liquids or 3 tobacco sticks, depending on the allocated arm). Participants randomized in the IQOS arm will receive one iQOS kit and a full 1 week supply of tobacco sticks of their choice (they will receive a number of tobacco sticks/day corresponding to the number of cigarettes smoked at baseline); those randomized in the JustFog-EC arm of the study will receive one JustFog Starter Kit and a full 1 week supply of e-liquids of their choice (they will receive 4, 10 mls refill containers).Free products will be supplied at each subsequent visit throughout the study. No supply of tobacco stick or e-liquid will be given at week-12, but users will be offered to keep using their products to minimize the risk of relapsing back to cigarette smoking. A prospective evaluation of cigarette consumption, adoption rates, acceptability and tolerability will be recorded throughout the study.

Visit 2 (V2):This will be scheduled 1 week after V1 (with a tolerance of +/- 3 days). Cigarette/day, eCO, AEs, BP, HR will be measured and product use recorded. Full 1 week supply of the chosen product will be provided.

Visit 3 (V3):This will be scheduled 2 weeks after V1 (with a tolerance of +/- 3 days). Cigarette/day, eCO, AEs, BP, HR will be measured and product use recorded. Participants will be instructed on how to collect and store their second urine sample before bringing it to the hospital at V4. Full 2 weeks supply of the chosen product will be provided.

Visit 4 (V4):This will be scheduled 4 weeks after V1 (with a tolerance of +/- 3 days). Cigarette/day, eCO, AEs, BP, HR will be measured, questionnaires completed and product use recorded. Step test will be carried out. Second urine sample will be collected, aliquotted and stored. Full 4 weeks supply of the chosen product will be provided.

Visit 5 (V5):This will be scheduled 8 weeks after V1 (with a tolerance of +/- 7 days). Cigarette/day, eCO, AEs, BP, HR will be measured, questionnaires completed and product use recorded. Full 4 weeks supply of the chosen product will be provided.

Visit 6 (V6):This will be scheduled 12 weeks after V1 (with a tolerance of +/- 7 days). Cigarette/day, eCO, AEs, BP, HR, weight, height will be measured, questionnaires completed and product use recorded. Step test will be carried out. No more products will be dispensed.

Follow-up Visit (V7):This final visit will be scheduled 24 weeks after V1 (with a tolerance of +/- 7 days)to review product usage and smoking behavior under naturalistic condition of use. Cigarette/day, eCO, AEs, BP, HR, weight, height will be measured, questionnaires completed and product use recorded. Step test will be carried out.

Data will be recorded from every subject on an electronic CRF, provided by a CRO, GCP compliant, 21 CFR Part 11 FDA compliant, listed in AIFA list of operating CRO. Urine samples will be collected at baseline and wk 4, and sent to an external laboratory for analytical assessment of selected Biomarkers of Exposure (BoE).

The study will be conducted at the University of Catania, Catania, Italy.

Participants Healthy smokers, not motivated to quit, will be randomized in two intervention groups in a 1:1 ratio to compare HTPs vs ECs in terms of reductions in cigarette consumption, adoption rate and acceptability, tolerability, and tobacco harm reduction. Sample size determination (better detailed below, in the relevant section) for no-inferiority testing is based on the assumptions that 1) expected quit rates based on most recent EC literature is about 20-25% and 2) that differences in quit rates between products under investigation should not exceed 10-15% (as per non-inferiority definition). According to these hypotheses the required number of participants per study arm is 104. Hence investigators intend to include 220 participants, 110 per group.

Study Products Tested

* Heated Tobacco Product (HTP):Investigators will use a HTP that does not involve combustion, generating a nicotine-containing aerosol. At the time of writing, IQOS is the only HTP available on the Italian market. IQOS is composed by: 1) a tobacco stick - a novel patent-pending tobacco product with unique processed tobacco made from tobacco powder; 2) an electronic holder into which the tobacco stick is inserted and which heats the tobacco by means of an electronically controlled heating blade; 3) a charger that is used to recharge the holder after each use.
* Investigators will use the three types of tobacco sticks specifically designed for IQOS(named HEETS) that are currently for sale in the Italian market: Heets Amber, Heets Yellow, and Heets Turquoise. These products are compliant to the EU Tobacco Product Directive.
* Electronic Cigarette (EC):JustFog Q16 Starter Kit and three types of e-liquid flavours, Puff Riserva Country 16 mg, Puff Riserva Toscana 16 mg, and Puff Artic 16 mg (2 tobacco-flavours and one menthol flavour), were chosen for the study.
* Products were selected by an Italian expert panel of 3 e-liquid producers and 3 vaping product distributors, moderated by the editor of a popular e-cigarette blog. Experts convened in Verona (Italy) during a major vaping expo event. Through consensus, the expert panel provided specific recommendation on the device(JustFog Q16 Starter Kit is one of the most popular e-cigarette device in Italy due to its good performance and quality, affordable price, and user friendliness especially for beginners) and the choice of e-liquids that could best match the sensorial experience of the iQOS tobacco sticks to be used in a switching study and minimize the local irritant effects of excessive PG/VG ratio. These products are compliant to the EU Tobacco Product Directive.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrolment into the study:

1. Able to comply with the study procedures
2. Male or female healthy smokers aged ≥19
3. Smoking at least 10 cigarettes a day
4. Smoking for at least one year
5. Not currently attempting to quit smoking or wishing to do so in the next 30 days (this will be verified at screening by the answer ''NO'' to both questions ''Do you intend to quit in the next 30 days?'' and ''Are you interested in taking part in one of our smoking cessation programs?'')
6. Female smokers not planning to become pregnant are using an acceptable form of contraception.

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrolment:

1. Use of smokeless tobacco, or any other tobacco products (including e-cigarettes, cigars, chewing tobacco, snus, etc.) within the last 3 months, at baseline and during the whole study.
2. Use of nicotine replacement therapy or other smoking cessation therapies within the last 3 months and at baseline.
3. Self-reported pregnancy, planned pregnancy or breastfeeding.
4. Tobacco industry employees and 1st degree relatives will be excluded in order to safeguard independence of the study

   -

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2019-05-25 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Catania, Italy, Catania, Italy

REFERENCES:
- [Derived] Caponnetto P, Campagna D, Maglia M, Benfatto F, Emma R, Caruso M, Caci G, Busa B, Pennisi A, Ceracchi M, Migliore M, Signorelli M. Comparing the Effectiveness, Tolerability, and Acceptability of Heated Tobacco Products and Refillable Electronic Cigarettes for Cigarette Substitution (CEASEFIRE): Randomized Controlled Trial. JMIR Public Health Surveill. 2023 Apr 4;9:e42628. doi: 10.2196/42628. PMID 37014673
- [Derived] Caponnetto P, Caruso M, Maglia M, Emma R, Saitta D, Busa B, Polosa R, Prosperini U, Pennisi A, Benfatto F, Sartorio C, Guastella M, Mondati E. Non-inferiority trial comparing cigarette consumption, adoption rates, acceptability, tolerability, and tobacco harm reduction potential in smokers switching to Heated Tobacco Products or electronic cigarettes: Study protocol for a randomized controlled trial. Contemp Clin Trials Commun. 2020 Jan 8;17:100518. doi: 10.1016/j.conctc.2020.100518. eCollection 2020 Mar. PMID 31956726

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IQOS | E-CIG
Started | 110 | 110
Completed | 110 | 101
Not Completed | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IQOS | E-CIG | Total
Number analyzed (Participants) | 110 | 110 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (16.1) | 41.3 (16.9) | 41.3 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 40 | 94
  Male | 56 | 70 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 110 | 110 | 220
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Smoking Cessation
Description: to compare the efficacy of HTP and EC, in terms of quit rates at week 12, by self-reporting abstinence from classic cigarette [validated by an Exhaled breath Carbon monoxide (eCO) measurement ≤10ppm)]
Time Frame: 12 WEEK
Measure: Count of Participants; unit: Participants
Arm/Group | IQOS | E-CIG
Number analyzed (Participants) | 110 | 107
Participants | 60 | 44
Statistical Analysis 1: Comparison: IQOS vs E-CIG; H0: P1-P2 ≤ -Margin; Test type: Non-Inferiority — Margin=0.04; p = 0.0051, Chi-squared, Corrected; Proportion Difference = 0.1342, 95% CI 2-sided [0.0014 to 0.2671]

2. Secondary Outcome: Number of Participants Smoking Reduction
Description: To compare the smoking reduction derived from the use of HTP and EC, intended as a 50% reduction in the number of conventional cigarette/day at week 12, defined through self-reporting;
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | IQOS | E-CIG
Number analyzed (Participants) | 110 | 107
Participants | 100 | 77
Statistical Analysis 1: Comparison: IQOS vs E-CIG; Test type: Superiority; p = 0.0003, Fisher Exact

3. Secondary Outcome: Adoption Rate
Description: To compare the adoption rate to product use [by collecting (empty) refill bottles and used heathsticks on a daily basis, verified by a study diary filled daily by the subject];
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Groups:
- IQOS: 4 PARTICIPANTS WITHOUT ADHERENCE IN IQOS GROUP
- E-CIG: 19 PARTICIPANTS WITHOUT ADHERENCE IN E-CIG GROUP
Arm/Group | IQOS | E-CIG
Number analyzed (Participants) | 110 | 107
Participants | 102 | 84
Statistical Analysis 1: Comparison: IQOS vs E-CIG; Test type: Superiority; p = 0.0003, Chi-squared, Corrected; Percentage Difference = 14.2

4. Secondary Outcome: Acceptability
Description: To compare the acceptability derived from the use of HTP and EC by the modified Cigarette Evaluation Questionnaire (mCEQ). It is a self-administered questionnaire that contains 12 items covering both reinforcing and aversive effects of smoking. The items are rated on a 7-point scale from 1 not at all to 7 extremely
  The total mCEQ score range from min 12 to max 84. Higher scores for the total mCEQ reflect a better outcome. There are also the following 5 subscales:
  1. Smoking Satisfaction (items 1, 2, 12) range of scores min 3 max 21;higher scores mean a better outcome.
  2. Psychological Reward (items 4-8), range of scores min 5 max 35; higher scores mean a better outcome.
  3. Aversion (items 9 and 10), range of scores min 2 max 14;higher scores mean a worse outcome.
  4. Single item score Enjoyment Respiratory Tract Sensations (item 3) range scores min 1 max 7;higher scores mean a better outcome.
  5. Single item score Craving Reduction (item 11), higher scores mean a better outcome
Time Frame: Week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- IQOS: MEAN CHANGES AT FINAL VISIT (WEEK 12) FROM BASELINE IN MCEQ SCORES: O.73
- E-CIG: MEAN CHANGES AT FINAL VISIT (WEEK 12) FROM BASELINE IN MCEQ SCORES: -O.17
Arm/Group | IQOS | E-CIG
Number analyzed (Participants) | 110 | 107
score on a scale | 0.73 [-1.04 to 2.49] | -0.17 [-1.77 to 1.44]

5. Secondary Outcome: Number of Participants With Product-related Adverse Events
Description: To compare number of participants with adverse events derived from the use of HTP and EC as assessed by CTCAE v4.0
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | IQOS | E-CIG
Number analyzed (Participants) | 110 | 110
Participants | 20 | 24

6. Secondary Outcome: Changes in Biomarkers of Biological Effects (BoBE)
Description: changes in Biomarkers of Biological Effects (BoBE) such as: eCO in the exhaled breath (i.e. eCO), step test values
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: ppm
Groups:
- IQOS: at v6 (week 12) mean(sd) eCO: 8.2 (8.0)
  at v6 (week 12) mean(sd) Step Test VoMax: 44.7 (28.7)
- E-CIG: at v6 (week 12) mean(sd) eCO: 10.1 (11.3)
  at v6 (week 12) mean(sd) Step Test VoMax: 50.9 (31.9)
Arm/Group | IQOS | E-CIG
Number analyzed (Participants) | 110 | 107
ppm | 8.2 (8.0) | 10.1 (11.3)

7. Secondary Outcome: Reliability
Description: To compare the reliability of HTP and EC, in terms of incidence and kind of malfunctioning events, through self-reporting.
Time Frame: Baseline visit, Week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Description: Any participants showed/reported signs and symptoms considered serious by the medical investigators with absence of all-cause of mortality
Arm/Group | IQOS | E-CIG
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/110
Other Adverse Events (participants affected / at risk) | 65/110 | 56/110
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IQOS (N=110) | E-CIG (N=110)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (27) | 24 (24)
Fatigue (General disorders) | 21 (21) | 12 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 15 (15)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7)
Palpitations (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT03569748/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT03569748/SAP_001.pdf